CLINICAL TRIAL: NCT00122642
Title: Short Daily Alcohol Locks for the Prevention of Tunneled Catheter Infection in Patients With Haematological Disease. Randomised Placebo Controlled Trial
Brief Title: Alcohol Locks for the Prevention of Tunneled Catheter-related Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Stichting Nuts Ohra (Other)
Responsible Party: BJ, Rijnders
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AL-01; SNO-T-07-57
Record Dates: First submitted 2005-07-19; First posted 2005-07-22 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Bacteremia
Keywords: catheterization; Catheters, Indwelling
MeSH Terms: conditions — Bacteremia | interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): The intervention is the instillation of ethanol 70% solution in the catheter lumen (or lumina) for 15minutes per day during hospital stay and for 15minutes for patients not in the hospital.
  Interventions: Procedure: Alcohol-lock
- 2 (Placebo Comparator): The intervention is the instillation of placebo solution in the catheter lumen (or lumina) for 15minutes per day during hospital stay and for 15minutes per week for patients not in the hospital.
  Interventions: Drug: placebo-lock

INTERVENTIONS:
Procedure: Alcohol-lock — The intervention is the instillation of ethanol 70% solution in the catheter lumen (or lumina) for 15minutes per day during hospital stay and for 15minutes per week for patients not in the hospital.
  Arms: 1
Drug: placebo-lock — The intervention is the instillation of placebo solution in the catheter lumen (or lumina) for 15minutes per day during hospital stay and for 15minutes per week for patients not in the hospital.
  Arms: 2

SUMMARY:
In modern-day medicine, the use of central venous catheters has become unavoidable. However, their use does not come without risk. It puts patients in danger of infectious complications (catheter-related infections [CRI]), the most important of which is catheter-related bloodstream infection (CRBSI). CRBSI is associated with a significant increase in hospital stay and, therefore, cost of patient management, morbidity, and probably also mortality. There still is an urgent need for effective, cheap and easy to implement measures to prevent CRI that are without risk of developing antibiotic resistance.

During use, bacteria can colonize the inner surface of the catheter. This endoluminal route of infection can be prevented to some extent when an antibiotic solution is instilled in the catheter for a long enough time and on a regular basis. However, to avoid resistance from occurring, the use of antibiotics for infection prevention should remain exceptional.

The use of a non-toxic antiseptic might be a better alternative. Recently, the use of an alcohol lock solution was suggested as a promising way to prevent CRBSI and the compatibility of polyurethane and silicone catheters submerged in an alcohol solution was publicized with no biomechanical or structural changes detected after 9 weeks of immersion. The major advantage of an alcohol lock solution would be the broad antimicrobial spectrum without the risk of compromising future antibiotic treatment as, in contrast to the use of an antibiotic lock, the development of antibiotic resistance is not of concern. Furthermore it would be cheap and universally available.

In this randomised study, the efficacy of a 70% alcohol lock solution for the prevention of CRBSI will be compared with placebo when applied for 15 minutes per day.

DETAILED DESCRIPTION:
In modern-day medicine, the use of intravascular catheters has become unavoidable. In the United States, hospitals and clinics purchase more than 150 million intravascular devices each year of which more than 5 million are central venous catheters. However, their use does not come without risk. It puts patients in danger of mechanical, thrombotic and infectious complications (catheter-related infections [CRI]), the most important of which is catheter-related bloodstream infection (CRBSI). CRBSI is associated with a significant increase in hospital stay and, therefore, cost of patient management, morbidity and probably also mortality. The increase in expenses was estimated to be 15,965 US dollars per patient with a CRBSI in 1994 and even 56,167 US dollars in another more recent study.

It is clear that the prevention of CRI is of utmost importance and will help to decrease patient suffering as well as cost of patient management. Extensive and detailed evidence-based recommendations for the prevention of CRI were recently published. However, many topics remain unresolved and there still is an urgent need for effective, cheap and easy to implement preventive measures that are without risk of developing antibiotic resistance.

Catheters can become colonized with microorganisms through exoluminal (catheter insertion site) or endoluminal (hub and infusates) routes. It has been shown that, the longer a catheter remains in place, the more important the endoluminal route becomes. The endoluminal route of infection can be prevented to some extent when an antibiotic solution is instilled in the catheter for a long enough time and on a regular basis. However, to avoid resistance from occurring, the use of antibiotics in such a lock for infection prevention should remain exceptional. Although there is evidence to support the concept, methodologically appropriate clinical data on the use of antiseptic solutions for this purpose are still awaited.

Recently, the use of an alcohol lock solution was suggested as a promising way to prevent CRBSI and the compatibility of polyurethane and silicone catheters submerged in an alcohol solution was publicized with no biomechanical or structural changes detected after 9 weeks of immersion. The major advantage of an alcohol lock solution would be the broad antimicrobial spectrum without the risk of compromising future antibiotic treatment as, in contrast to the use of an antibiotic lock, the development of antibiotic resistance is not of concern. Furthermore it would be cheap and universally available.

In this randomised study the efficacy of a 70% alcohol lock solution for the prevention of CRBSI will be compared with placebo when applied for 15 minutes per day.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old
* Admitted to the haematology department
* Had a tunnelled central venous catheter inserted in the preceding 72 hours

Exclusion Criteria:

* Known allergy to alcohol or active use of metronidazole (or related 2-nitroimidazole compounds) or disulfiram (Antabuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2005-08; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Endoluminal catheter related bacteremia | at time of catheter removal

SECONDARY OUTCOMES:
All catheter-related bacteremias with differential time to positivity (DTTP) > 2 hours | at time of catheter removal
Catheter survival time | at time of catheter removal
Vancomycin and linezolid use | at time of catheter removal
Incidence of positive catheter tip cultures | at time of catheter removal
Incidence of bacteremia/fungemia (catheter-related or not) | at time of catheter removal

CONTACTS AND LOCATIONS:
Overall Officials: Bart JA Rijnders, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Background] Mermel LA, Farr BM, Sherertz RJ, Raad II, O'Grady N, Harris JS, Craven DE; Infectious Diseases Society of America; American College of Critical Care Medicine; Society for Healthcare Epidemiology of America. Guidelines for the management of intravascular catheter-related infections. Clin Infect Dis. 2001 May 1;32(9):1249-72. doi: 10.1086/320001. Epub 2001 Apr 3. No abstract available. PMID 11303260
- [Background] Digiovine B, Chenoweth C, Watts C, Higgins M. The attributable mortality and costs of primary nosocomial bloodstream infections in the intensive care unit. Am J Respir Crit Care Med. 1999 Sep;160(3):976-81. doi: 10.1164/ajrccm.160.3.9808145. PMID 10471627
- [Background] Rello J, Ochagavia A, Sabanes E, Roque M, Mariscal D, Reynaga E, Valles J. Evaluation of outcome of intravenous catheter-related infections in critically ill patients. Am J Respir Crit Care Med. 2000 Sep;162(3 Pt 1):1027-30. doi: 10.1164/ajrccm.162.3.9911093. PMID 10988125
- [Background] Renaud B, Brun-Buisson C; ICU-Bacteremia Study Group. Outcomes of primary and catheter-related bacteremia. A cohort and case-control study in critically ill patients. Am J Respir Crit Care Med. 2001 Jun;163(7):1584-90. doi: 10.1164/ajrccm.163.7.9912080. PMID 11401878
- [Background] Dimick JB, Pelz RK, Consunji R, Swoboda SM, Hendrix CW, Lipsett PA. Increased resource use associated with catheter-related bloodstream infection in the surgical intensive care unit. Arch Surg. 2001 Feb;136(2):229-34. doi: 10.1001/archsurg.136.2.229. PMID 11177147
- [Background] O'Grady NP, Alexander M, Dellinger EP, Gerberding JL, Heard SO, Maki DG, Masur H, McCormick RD, Mermel LA, Pearson ML, Raad II, Randolph A, Weinstein RA. Guidelines for the prevention of intravascular catheter-related infections. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 Aug 9;51(RR-10):1-29. PMID 12233868
- [Background] Raad I, Costerton W, Sabharwal U, Sacilowski M, Anaissie E, Bodey GP. Ultrastructural analysis of indwelling vascular catheters: a quantitative relationship between luminal colonization and duration of placement. J Infect Dis. 1993 Aug;168(2):400-7. doi: 10.1093/infdis/168.2.400. PMID 8335977
- [Background] Carratala J, Niubo J, Fernandez-Sevilla A, Juve E, Castellsague X, Berlanga J, Linares J, Gudiol F. Randomized, double-blind trial of an antibiotic-lock technique for prevention of gram-positive central venous catheter-related infection in neutropenic patients with cancer. Antimicrob Agents Chemother. 1999 Sep;43(9):2200-4. doi: 10.1128/AAC.43.9.2200. PMID 10471564
- [Background] Schwartz C, Henrickson KJ, Roghmann K, Powell K. Prevention of bacteremia attributed to luminal colonization of tunneled central venous catheters with vancomycin-susceptible organisms. J Clin Oncol. 1990 Sep;8(9):1591-7. doi: 10.1200/JCO.1990.8.9.1591. PMID 2202792
- [Background] Dogra GK, Herson H, Hutchison B, Irish AB, Heath CH, Golledge C, Luxton G, Moody H. Prevention of tunneled hemodialysis catheter-related infections using catheter-restricted filling with gentamicin and citrate: a randomized controlled study. J Am Soc Nephrol. 2002 Aug;13(8):2133-9. doi: 10.1097/01.asn.0000022890.29656.22. PMID 12138146
- [Background] Henrickson KJ, Axtell RA, Hoover SM, Kuhn SM, Pritchett J, Kehl SC, Klein JP. Prevention of central venous catheter-related infections and thrombotic events in immunocompromised children by the use of vancomycin/ciprofloxacin/heparin flush solution: A randomized, multicenter, double-blind trial. J Clin Oncol. 2000 Mar;18(6):1269-78. doi: 10.1200/JCO.2000.18.6.1269. PMID 10715297
- [Background] Chatzinikolaou I, Zipf TF, Hanna H, Umphrey J, Roberts WM, Sherertz R, Hachem R, Raad I. Minocycline-ethylenediaminetetraacetate lock solution for the prevention of implantable port infections in children with cancer. Clin Infect Dis. 2003 Jan 1;36(1):116-9. doi: 10.1086/344952. Epub 2002 Dec 11. PMID 12491212
- [Background] Allon M. Prophylaxis against dialysis catheter-related bacteremia with a novel antimicrobial lock solution. Clin Infect Dis. 2003 Jun 15;36(12):1539-44. doi: 10.1086/375234. Epub 2003 Jun 6. PMID 12802753
- [Background] Maki DG, Crnich CJ, Safdar N. Successful use of a 25% Alcohol Lock Solution for Prevention of Recurrent CVC-Related Bloodstream Infection in a patient on Home TNA. 42nd ICAAC Abstracts, American Society for Microbiology, September 27 - 30, 2002, San Diego, CA, page 320 . 2002.
- [Background] A.Aiyangar, W.C.Crone, C.J.Crnich DGM. Effect of Ethanol on the Mechanical Properties of Polyurethane Catheters. Proceedings of the 2002 SEM Annual Conference and Exposition on Experimental and Applied Mechanics . 2002.
- [Derived] Slobbe L, Doorduijn JK, Lugtenburg PJ, El Barzouhi A, Boersma E, van Leeuwen WB, Rijnders BJ. Prevention of catheter-related bacteremia with a daily ethanol lock in patients with tunnelled catheters: a randomized, placebo-controlled trial. PLoS One. 2010 May 26;5(5):e10840. doi: 10.1371/journal.pone.0010840. PMID 20520776